CLINICAL TRIAL: NCT02987205
Title: A Multicenter, Double-Blind, Randomized, Split-Face Study to Evaluate the Safety and Efficacy of Revanesse® Ultra Versus Restylane® for the Correction of Nasolabial Folds
Brief Title: Multicenter Double-Blind Randomized Split-Face Study to Evaluate Revanesse® Ultra vs Restylane® for Correction of NLF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prollenium Medical Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SYM2014-02
Record Dates: First submitted 2016-12-05; First posted 2016-12-08 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2017-11

CONDITIONS: Nasolabial Fold Correction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

ARMS (2):
- Revanesse Ultra (Experimental): Revanesse Ultra in the NLF on one side of the face
  Interventions: Device: Revanesse Ultra
- Restylane (Active Comparator): Restylane injection in the NLF on the other side of the face to optimal correction
  Interventions: Device: Restylane

INTERVENTIONS:
Device: Revanesse Ultra — NLF correction
  Arms: Revanesse Ultra
Device: Restylane — NLF Correction
  Arms: Restylane

SUMMARY:
A randomized, multicenter, double blind, split-face study in subjects seeking NLF correction. Subjects were treated with Revanesse Ultra in the NLF on one side of the face and Restylane in the NLF on the other side of the face. The side of the face for each product was randomly assigned. The investigator performing the evaluations and the subject were blinded to the treatment; injections of the study product were performed by an unblinded injecting investigator.

DETAILED DESCRIPTION:
The study was a randomized, double-blind prospective, comparative study of the efficacy and safety of Revanesse Ultra versus the approved product Restylane in the cutaneous correction of NLFs. Randomization followed a 1:1 within-subject control model of augmentation correction of NLFs. Given that the implants have been shown to not migrate, the within-subject model was ideal and had already been shown in previous studies to detect differences. Subjects with signs of NLFs who met the entry criteria were enrolled. All subjects were followed for efficacy and safety for 6 months. Subjects could have open-label retreatment as needed with Revanesse Ultra at 6 months if their baseline WSRS scores had returned to baseline, or as needed to achieve optimal correction if their baseline WSRS scores had not returned to baseline and were followed for a total of 12 months. The study design was appropriate for the indication studied.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be eligible for the study:

1. Men or women 22 years of age or older.
2. Two fully visible bilateral nasolabial folds each with a Wrinkle Severity Rating Scale Score of 3 or 4 that may be corrected with an injectable dermal filler.
3. If female and of childbearing potential, a negative urine pregnancy test and agree to use adequate contraception. Female subjects of childbearing potential (excluding women who are surgically sterilized or postmenopausal for at least 2 years) must have a negative urine pregnancy test and must be willing to use a medically accepted method of contraception during the study. The following are considered acceptable methods of birth control for the purpose of this study: oral contraceptives, contraceptive patches, contraceptive implant, vaginal contraceptive, double barrier methods (e.g., condom and spermicide), contraceptive injection (Depo-Provera®), intrauterine device (IUD), hormonal IUD (Mirena®), and abstinence with a documented second acceptable method of birth control if the subject becomes sexually active. Subjects entering the study who are on hormonal contraceptives must have been on the method for at least 90 days prior to the study and continue the method for the duration of the study. Subjects who had used hormonal contraception and stopped must have stopped no less than 90 days prior to Visit 1/Day 1.
4. Ability to understand and comply with the requirements of the study.
5. Willingness and ability to provide written informed consent.
6. Agree to refrain from seeking other treatment for this condition during the study.

   -

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study:

1. Wrinkle Severity Rating Scale Score of ≤ 2 on the right or left nasolabial fold.
2. Women who are pregnant or lactating.
3. Received prior dermabrasion, facelift, or Botox below the orbital rim within 6 months (180 days) prior to entry into the study.
4. Previous tissue augmentation (bulking agents) for facial wrinkles and scars within 6 months (180 days) at the proposed injection sites.
5. Previous tissue augmentation with permanent implants.
6. Evidence of scar-related disease or delayed healing activity within the past 1 year.
7. Scars at the intended treatment sites.
8. History of keloid formation or hypertrophic scars.
9. Any infection or wound on the face.
10. Allergic history including anaphylaxis or multiple severe allergies to natural rubber latex or lidocaine.
11. Aspirin or nonsteroidal anti-inflammatory drugs within 1 week (7 days) prior to treatment.
12. Concomitant anticoagulant therapy, antiplatelet therapy, or history of bleeding disorders or connective tissue disorders.
13. Over-the-counter (OTC) wrinkle products or prescription wrinkle treatments within 4 weeks (28 days) prior to treatment and throughout the study.
14. Immunocompromised or immunosuppressed.
15. Clinically significant organic disease including clinically significant cardiovascular, hepatic, pulmonary, neurologic, or renal disease or other medical condition, serious intercurrent illness, or extenuating circumstance that, in the opinion of the investigator, preclude participation in the trial.
16. Received any investigational product within 30 days of signing the Informed Consent Form.
17. Facial tattoo that may interfere with diagnosis.
18. Systemic (oral/injectable) corticosteroids or immunosuppressive medications within 30 days prior to treatment and topical steroids on the face within 14 days prior to treatment start and throughout the study.

    -

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2015-05; Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Gold, MD, Principal Investigator — Tennessee Clinical Research Center

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Bilateral Treatment With Revanesse Ultra and Restylane: Randomized treatment with Revanesse Ultra in the Nasolabial Fold (NLF) on one side of the face, and Restylane on the opposite side of the face - the study is a randomized, multicenter, double blind, split-face study in subjects seeking NLF correction. Subjects were treated with Revanesse Ultra in the NLF on one side of the face and Restylane in the NLF on the other side of the face. The side of the face for each product was randomly assigned.
Period: Overall Study
Arm/Group | Bilateral Treatment With Revanesse Ultra and Restylane
Started | 163
Treated - Bilateral NLF Injection | 163
Completed | 159 (Treatment is bilateral, subject lost to Restylane AE was lost to further Revanesse Ultra treatment)
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: There were 163 participants enrolled and treated, the participants received bilateral NLF injection with Revanesse Ultra in one NLF, and Restylane in the other NLF
Units Other Than Participants: NLF Treatments
Groups:
- Split Face Study Bilateral Revanesse Ultra vs Restylane in NLF: Split face study - Revanesse Ultra in the NLF on one side of the face and Restylane on the opposite side of the face for NLF correction, treatment is randomized
Arm/Group | Split Face Study Bilateral Revanesse Ultra vs Restylane in NLF
Number analyzed (Participants) | 163
Number analyzed (NLF Treatments) | 326
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (10.16)
Age, Customized [Count of Participants; unit: Participants]
  22 to <40 years | 15
  40 to <64 years | 110
  64 to <75 years | 35
  = or >75 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 156
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 146
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 154
  More than one race | 1
  Unknown or Not Reported | 0
Fitzpatrick Skin Type (FST) Classification [Count of Participants; unit: Participants] — FST Type I skin always burns, never tans (pale white; blond or red hair; blue, gray eyes; freckles) FST Type II skin usually burns, tans minimally (white; blond, brown or red hair; blue, green, or hazel eyes) FST Type III skin sometimes has a mild burn, tans uniformly (cream white; yellowish; any hair color or brown eyes) FST Type IV skin burns minimally, always tans well (light brown; olive; dark brown to black hair) FST Type V skin very rarely burns, tans very easily (brown) FST Type VI skin never burns, always tans (deeply pigmented dark brown to darkest brown, black in complexion)
  Participants
    FST I | 3
    FST II | 50
    FST III | 83
    FST IV | 16
    FST V | 4
    FST VI | 7
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI is the body mass divided by the square of the body height, and is universally expressed in units of kg/m^2
  kg/m^2 | 26.27 (5.374)

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Variable is Change From Baseline to Visit 6/Week 24 in Wrinkle Severity Rating Scale (WSRS) Score
Description: Primary efficacy variable is change from Baseline to Visit 6/Week 24 in Wrinkle Severity Rating Scale (WSRS) - Treatment success is defined as at least a 1-grade improvement in WSRS from baseline to Week 24
  WSRS Score categories:
  1. Absent - No visible fold; continuous skin line.
  2. Mild - Shallow but visible fold with a slight indentation; minor facial feature; implant is expected to produce a slight improvement in appearance.
  3. Moderate - Moderately deep folds; clear facial feature visible at normal appearance but not when stretched; excellent correction is expected from injectable implant.
  4. Severe - Very long and deep folds; prominent facial feature; less than 2 mm visible when stretched; significant improvement is expected from injectable implant.
  5. Extreme - Extremely deep and long folds, detrimental to facial appearance; 2 to 4 mm visible V-shaped fold when stretched; unlikely to have satisfactory correction with injectable implant alone.
Time Frame: Visit 6/Week 24
Population: Analysis of effectiveness based on Per Protocol analysis which includes 125 evaluable patients at 24 weeks.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Units Other Than Participants: Nasolabial Folds
Arm/Group | Revanesse Ultra | Restylane
Number analyzed (Participants) | 125 | 125
Number analyzed (Nasolabial Folds) | 125 | 125
scores on a scale | 1.02 [0.902 to 1.146] | 0.91 [0.777 to 1.047]
Statistical Analysis 1: Comparison: Revanesse Ultra vs Restylane; Test type: Non-Inferiority — If the upper bound of this 95% CI was less than the prespecified non-inferiority limit of 0.50, the Test product would be claimed to be non-inferior to the Comparator product; p = 0.0130, Wilcoxon (Mann-Whitney) — Wilcoxon matched-pairs signed rank test

2. Secondary Outcome: Secondary Efficacy Endpoints Are the Responder Rate, Percentage of *Nasolabial Folds* With Treatment Success
Description: Treatment success (defined as at least a 1-grade improvement in WSRS from baseline to Week 24):
  The WSRS Score is a 5-point scale. The WSRS score was assessed for each NLF at every study visit through Visit 6/Week 24 by a blinded evaluator (blinded to the treatment assignment of each NLF).
Time Frame: Visit 6/Week 24
Population: Per-Protocol (PP) Population
Measure: Count of Units; unit: Nasolabial Folds
Units Other Than Participants: Nasolabial Folds
Arm/Group | Revanesse Ultra | Restylane
Number analyzed (Participants) | 125 | 125
Number analyzed (Nasolabial Folds) | 125 | 125
Nasolabial Folds | 98 | 91

3. Other Pre Specified Outcome: Other Efficacy Variables Include Change in WSRS Score
Description: Treatment success is (defined as at least a 1-grade improvement in WSRS from baseline to Week 24)
Time Frame: Visit 2/Week 1, Visit 3/Week 2, Visit 4/Week 4, and Visit 5/Week 12
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Other Efficacy Variables Include Change in Patient Global Aesthetic Improvement (pGAI) Score
Description: Treatment success is (defined as at least a 1-grade improvement in WSRS from baseline to Week 24)
Time Frame: Visit 2/Week 1, Visit 3/Week 2, Visit 4/Week 4, and Visit 5/Week 12
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Other Efficacy Variables Include Change in Investigator Global Aesthetic Improvement (iGAI) Score
Description: Treatment success is (defined as at least a 1-grade improvement in WSRS from baseline to Week 24)
Time Frame: Visit 2/Week 1, Visit 3/Week 2, Visit 4/Week 4, and Visit 5/Week 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Treatment safety was evaluated by frequency and percent of subjects and investigators reporting treatment-emergent adverse events (TEAEs) tabulated by treatment group, location, frequency, severity and duration after each treatment (initial treatment, touch up) and throughout the study. TEAEs were assessed by a subject diary after each injection, touch up and follow up visit, and were reported by the Evaluating Investigator at each of the follow-up visits
Arm/Group | Revanesse Ultra | Restylane
All-Cause Mortality (participants affected / at risk) | 0/163 | 0/163
Serious Adverse Events (participants affected / at risk) | 0/163 | 1/163
Other Adverse Events (participants affected / at risk) | 114/163 | 137/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Revanesse Ultra (N=163) | Restylane (N=163)
Treatment emergent Injection site vascular complication (General disorders) | 0 (0) | 1 (1) — Device related serious adverse event of a possible vascular event
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Revanesse Ultra (N=163) | Restylane (N=163)
INJECTION SITE HAEMATOMA (General disorders) | 82 (106) | 77 (95) — bruising at the injection site
INJECTION SITE SWELLING (General disorders) | 77 (102) | 116 (163) — swelling at the injection site
INJECTION SITE PAIN (General disorders) | 62 (103) | 108 (192) — pain at the injection site
INJECTION SITE ERYTHEMA (General disorders) | 35 (44) | 52 (65) — redness at the injection site

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There are restrictions within the site contracts that the sites cannot publish any results and also have confidentiality agreements in place separately that restrict any publications by sites regarding results, findings, etc.

DOCUMENTS (1):
  • Study Protocol (2015-10-28): https://cdn.clinicaltrials.gov/large-docs/05/NCT02987205/Prot_000.pdf